CLINICAL TRIAL: NCT07135154
Title: Comparison of Balanced Anesthesia Protocols in Gastric Sleeve Surgery in Terms of Postoperative Opioid Consumption
Brief Title: Postoperative Opioid Consumption in Gastric Sleeve Surgery
Acronym: POCiGSS
Status: Active, not recruiting | Type: Observational
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Serkan Uckun, assistant professor, Balikesir University
Other Study IDs: 2025/275
Record Dates: First submitted 2025-08-13; First posted 2025-08-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Obesity &Amp; Overweight; General Anesthetic; Ketamine
Keywords: obesity; general anesthesia; ketamine
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fentanyl: Fentanyl
- Fentanyl+Ketamine: Ketamine

SUMMARY:
The study aimed to compare balanced anesthesia protocols using only opioids as analgesics during induction in gastric sleeve surgery with protocols using opioids and ketamine together in terms of anesthesia management, opioid side effects, and postoperative analgesia.

DETAILED DESCRIPTION:
During gastric sleeve surgery under general anesthesia, various drugs are administered intraoperatively to induce loss of consciousness, immobility, and pain relief (analgesia). Opioids are the most commonly used analgesics. However, the response to opioids varies widely, and their use is associated with significant side effects. In balanced general anesthesia, in addition to opioid medications, hypnotics, NMDA antagonists (ketamine, magnesium sulfate), sodium channel blockers (local anesthetics), anti-inflammatory drugs (NSAIDs, dexamethasone), and alpha-2 agonists (dexmedetomidine, clonidine) may be used. One of the components of ERAS (Enhanced Recovery After Surgery) protocols, which aim to reduce metabolic stress developing in response to surgery and promote rapid recovery after surgery, is to provide effective postoperative analgesia while using opioids as little as possible. These different anesthesia approaches may offer options for surgery.

The addition of ketamine to anesthesia induction and maintenance may affect postoperative opioid consumption. Adding ketamine to anesthesia induction and maintenance may affect postoperative opioid consumption. Reducing opioid consumption can prevent opioid-related side effects such as nausea, constipation, and itching.

Opioid-related side effects such as nausea, constipation, and itching can be prevented by reducing opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

Patients who have undergone gastric sleeve surgery Patients with mild systemic disease Patients with severe systemic disease that does not affect daily activities

Exclusion Criteria:

Those with data loss in their files Those who do not use patient-controlled analgesia devices Patients who did not undergo standard anesthesia protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who have undergone gastric sleeve surgery in the general surgery operating room at Balıkesir University Hospital
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-03-29 (Actual); Study Completion 2026-02-06 (Estimated)

PRIMARY OUTCOMES:
Morphine equivalent opioid consumption | 24 hours

SECONDARY OUTCOMES:
Postoperative pain | 24 hours
  Postoperative pain is assessed using a numerical pain scale. The Numerical Pain Rating Scale (NRS) was used in the study. NRS pain scores range from 0 (no pain) to 10 (most severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Balıkesir University Health Practice and Research Hospital, Balıkesir, Turkey (Türkiye)